CLINICAL TRIAL: NCT03462355
Title: Tobacco Smoking Among Crosslinked-keratoconus Patients
Acronym: TOBACOLINK
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-02Obs-CHRMT
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Certain studies reported that cigarette by-products may make the cornea more rigid, suggesting that it could lead to "natural" CXL of collagen fibers, hence a protective effect for KC. Others have reported that cigarette smoking causes no significant changes in the corneal biomechanics. The aim of this study was to assess a possible link between keratoconus (KC) occurrence and patients' smoking habits.

DETAILED DESCRIPTION:
a telephone Survey was performed among 80 KC patients who were treated from March 2014 until September 2017 by accelerated crosslinking (A-CXL) within the ophthalmology department. From the 80 people we phoned, 62 answered. Our questions were regarding family history, allergic history, and smoking habits. Family history was considered positive if a first-degree or second-degree relative had been diagnosed with KC. Allergies toward any kind of external factors were marked as positive. Patients' smoking habits were recorded and classified into regular, occasional, ex-smoker and non-smoker. The results were confronted to those of the general population by indirect standardization over age and sex according to the "Baromètre Santé 2010" INPES survey (French Nation Institute for Prevention and Health Education).

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from Keratoconus and needing Cross-linking therapy

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients suffering from Keratoconus and needing Cross-linking therapy
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Percentage of smokers | After 2 years
  Percentage of smokers among Cross-linked Keratoconus patients